CLINICAL TRIAL: NCT06314503
Title: Clinical Validation of a Continuous Flow Peritoneal Dialysis System With Dialysate Regeneration
Brief Title: First-in-human Study to Examine Safety of a New Peritoneal Dialysis Device (WEAKID) in End-stage Kidney Disease Patients
Acronym: CORDIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Horizon 2020 - European Commission (Other); Dutch Kidney Foundation (Other); Health Holland (Other); Nanodialysis Ltd (Unknown); University of Modena and Reggio Emilia (Other); Servicio Madrileno De Salud (SERMAS) (Unknown); PPI Healthcare Consulting Ltd (Unknown)
Responsible Party: Principal Investigator, Karin G.F. Gerritsen, MD, PhD, Associate professor, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-075_CORDIAL_FIH; NL83843.000.23 (Other: CCMO (Centrale Commissie Mensgebonden Onderzoek))
Record Dates: First submitted 2024-01-01; First posted 2024-03-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic; Chronic Kidney Diseases
Keywords: Peritoneal Dialysis; First-in-human; Medical device
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This study has a first-in-human, prospective, open-label, non-randomized, three-center, single-arm design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WEAKID (Experimental): Six treatments over the course of two weeks with the WEAKID system
  Interventions: Device: WEAKID

INTERVENTIONS:
Device: WEAKID — Six treatments over the course of two weeks with the WEAKID system:
  * Week 1 (without the sorbents)
    * Day 1: four-hour treatment
    * Day 2: eight-hour treatment
    * Day 3: eight-hour treatment
  * Week 2 (with the sorbents)
    * Day 1: four-hour treatment
    * Day 2: eight-hour treatment
    * Day 3: eight-hour treatment
  Other Names: CORDIAL

SUMMARY:
The goal of this first-in-human clinical trial is to examine the safety and efficacy of treatment with a new peritoneal dialysis (PD) device called WEAKID (WEarable Artificial KIDney for peritoneal dialysis). This device, unlike conventional PD, allows for continuous flow of dialysate inside the abdominal cavity combined with continuous regeneration of spent dialysate thanks to sorbents that remove toxins from the fluid.

The study will include PD patients of 18 years or older with a well-functioning peritoneal catheter and no history of a PD-related infection for at least eight weeks prior to enrolment.

The main purpose of this study is to assess the (short-term) safety of the WEAKID system in a limited number (n=12) of patients and sessions.

Participants will undergo six treatment sessions (of four or eight hours) in total over a period of two weeks, either with or without a sorbent chamber.

Participants will be asked to collect urine and dialysate the week before the first treatment and during the treatment days. In addition, blood samples will be collected before and during the treatment weeks in order to compare the effects of conventional PD with that of WEAKID treatment. A peritoneal equilibrium test will also be done before and after the treatment weeks to test the function of the lining of the abdomen (the peritoneal membrane).

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is a life-sustaining renal replacement therapy for patients with end-stage kidney disease (ESKD). With PD, waste solutes and excess water are drawn from the blood across the peritoneal membrane lining the abdominal cavity via diffusion and osmosis, respectively, into dialysis fluid (peritoneal dialysate) that is introduced into the abdominal cavity through a permanent tube (peritoneal catheter). The peritoneal dialysate is replaced 4-6 times/day either manually by the patient or automatically by a machine at night while the patient is asleep. PD is a gentle dialysis technique that provides continuous gradual dialysis while the patient is free to move during the day. However, PD has several disadvantages. Removal of waste solutes is inadequate and technique failure rate is high, contributing to poor quality of life and high (co)morbidity and mortality (10-15% per year). The low solute clearance (~1-7% of that of healthy kidneys (depending on the solute) and lower than that with haemodialysis (HD)) is due to rapid decrease of diffusive transport of solutes during a dwell due to the disappearance of the plasma-to-dialysate concentration gradient across the peritoneal membrane. The limited technique survival (median 3.7 years) is primarily due to the high incidence of recurrent infection of the peritoneal membrane (peritonitis) and exposure of the peritoneal membrane to very high, harmful glucose concentrations needed for osmotic fluid removal.

Both peritonitis and high glucose concentrations cause pathological changes of the peritoneal membrane and eventually ultrafiltration failure necessitating a switch to the more invasive and expensive HD treatment. To reduce the existing shortcomings of conventional PD, a novel continuous flow peritoneal dialysis system with dialysate regeneration (WEAKID) for PD was developed. WEAKID treatment is based on continuous recirculation of peritoneal dialysate via the single lumen peritoneal catheter with regeneration of spent dialysate by means of sorbent technology. The WEAKID nighttime system (weight: ~12 kg) is intended to be used for 8h per day (during the night) on a daily basis. Instead of performing 4-6 exchanges with fresh peritoneal dialysate per day, WEAKID uses one peritoneal dialysate filling which is continuously recirculated and regenerated. The continuous regeneration prevents saturation of the dialysate with toxins and thereby maintains a high plasma to dialysate concentration gradient which enhances diffusive transport of uremic toxins. In addition, the continuous recirculating flow of fluid along the peritoneal membrane is expected to increase the mass transfer area coefficient as observed in previous studies with continuous flow peritoneal dialysis, probably due to reduction of diffusion resistance, renewal of stagnant fluid layers at the tissue surface and an increase of the effective membrane area. Both the high plasma to dialysate concentration gradient and the increase in mass transfer contribute to an enhancement of the clearance. Another advantage of the WEAKID system is that the glucose peak load to peritoneum is lower than with traditional automated peritoneal dialysis (APD) and continuous ambulatory peritoneal dialysis (CAPD) thanks to the buffering of the sorbents (sorbents adsorb glucose at the start, lowering the initial glucose peak, and release the glucose again at later stage) and the continuous recirculation.

The primary objective of this study is to assess the (short-term) safety of the WEAKID nighttime system in a limited number (n=12) of patients and sessions (6 sessions per patient).

Secondary objectives of this study are:

1. To evaluate the incidence of adverse events (AEs) and device deficiencies (DDs) other than serious adverse device effects (SADEs) and DDs that could have led to a serious adverse event (SAE)
2. To describe the characteristics of WEAKID treatment (i.e. number and duration of sessions, dialysate flow rates)
3. To evaluate the clinical condition and vital signs of the participants during WEAKID treatment
4. To evaluate the effectiveness of ultrafiltration (UF) in relation to glucose concentration during WEAKID treatment
5. To evaluate the efficacy of solute removal and base release of WEAKID treatment
6. To evaluate the evolution of plasma analytes during WEAKID treatment
7. To evaluate the evolution of dialysate effluent analytes of the WEAKID system
8. To evaluate the (technical) device performance of the WEAKID system by the number of device deficiencies, adverse device effects and changes in intraperitoneal pressure
9. To evaluate patient tolerance during WEAKID treatment
10. To evaluate the evolution of uremic symptoms during WEAKID treatment
11. To evaluate the effectiveness of using sorbents for dialysate regeneration and the effectiveness of continuous recirculating flow in relation to the efficacy of solute removal.

The WEAKID system will be tested in a clinical setting on 6 days over a period of 2 weeks. During the first week, the subjects will be treated with the nighttime system without sorbents for 4h (first day) or 8h (second and third day) during daytime. The second week, treatment will consist of the nighttime system with sorbents (also 4h (first day) or 8h (second and third day) during daytime).

This way, exposure to new components of the system is incremental and the effectiveness of the sorbents can be analyzed separately from the effect of continuous recirculating flow dialysis. A peritoneal equilibration test (PET) will be performed at baseline and follow-up. In addition, patients will collect 24h spent peritoneal dialysate and 24h urine followed by venous puncture for blood sampling 3 times prior to WEAKID treatment during standard PD.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Treated with PD for at least 3 months prior to enrolment
* Well-functioning peritoneal catheter and no peritoneal catheter replacement for at least a month prior to enrolment
* No PD-related infection (exit-site infection, tunnel infection or peritonitis) less than 8 weeks prior to enrolment (counting from the day that the treatment has been finished).
* Previous or current use of Extraneal® with no contra-indications
* Capable of understanding the patient information sheet and informed consent form (ICF) and give informed consent
* Willing and able to comply with all study procedures and attend all study visits

Exclusion Criteria:

* Patients who are unable to provide informed consent
* Patients who are unable to comply with study procedures
* Patients who received renal replacement therapy other than conventional PD less than 8 weeks prior to enrolment
* Patients who participated in an intervention trial less than 8 weeks prior to enrolment or are currently participating in an intervention trial. Patients in an observational study without any interventions or in post-market surveillance do not need to be excluded.
* Patients with a PD-related infection (exit-site infection, tunnel infection or peritonitis) less than 8 weeks prior to enrolment (counting from the day that the treatment has been finished)
* Patients with peritoneal catheter dysfunction or mechanical issues less than one month prior to enrolment
* Patients who have never used Extraneal® dialysis fluid or have a contra-indication for Extraneal®: a known allergy to cornstarch or icodextrin; maltose or isomaltose intolerance; glycogen storage disease
* Patients with an incompatible PD connection to the device (e.g. Fresenius PD system)
* Patients with haemoglobin concentrations < 6.2 mmol/L (< 10 g/dL) less than 8 weeks prior to enrolment
* Patients with hyperkalemia (> 6.0 mmol/L) or hyponatremia (< 130 mmol/L) in the 8 weeks prior to enrolment
* Patients with hypocalcemia (plasma total calcium concentration corrected for albumin <2.20 mmol/L or ionized calcium <1.15 mmol/L) or hypomagnesemia (plasma magnesium concentration <0.70 mmol/L) in the 8 weeks prior to enrolment
* Patients with any serious medical condition which in the opinion of the investigator, may adversely affect the safety of the participant and/or effectiveness of the study
* Female patients who are either (planning to become) pregnant within the study period or breast feeding
* Patients with a life expectancy <3 months
* Anticipated living donor kidney transplantation <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serious adverse device effects (SADEs) and device deficiencies (DDs) | This will be assessed through study completion (four weeks in total per participant)
  Serious adverse device effects (SADEs) and device deficiencies (DDs) that could have led to a serious adverse event
Critical changes in blood pressure | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in blood pressure (measured in mmHg; both systolic and diastolic pressures will be assessed).
Critical changes in heart rate | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in heart rate (measured in beats per minute).
Critical changes in body temperature | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in body temperature (measured in °C).
Critical changes in oxygen saturation | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in oxygen saturation (measured in %).
Critical changes in plasma potassium | This will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in plasma potassium (before and after WEAKID treatment in mmol/L).
Critical changes in plasma calcium | This will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in plasma calcium (before and after WEAKID treatment in mmol/L).
Critical changes in plasma bicarbonate | This will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in plasma bicarbonate (before and after WEAKID treatment in mmol/L).
Critical changes in intra-abdominal dialysate volume | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in intra-abdominal dialysate volume.
Critical changes in intra-abdominal pressure | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Critical changes requiring intervention in intra-abdominal dialysate pressure (in mbar).

SECONDARY OUTCOMES:
Adverse events (AEs) and device deficiencies (DDs) | This will be assessed through study completion (four weeks in total per participant)
  Assessing incidence of adverse events (AEs) and device deficiencies (DDs) other than SADEs and DDs that could have led to an serious adverse event (SAE).
Number of WEAKID treatments | The number of WEAKID treatments will be assessed for the study treatment period (2 weeks in total per participant)
  The number of WEAKID treatments per patient will be determined
Duration of WEAKID treatments | This will be assessed for each WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Duration of each WEAKID treatment will be assessed (in minutes).
Dialysate flow rates during WEAKID treatment | This will be assessed during WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Dialysate flow rates will be determined during each WEAKID treatment (in mL/min).
Evolution of blood pressure | This will be assessed during WEAKID treatment at t=0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Blood pressure will be measured multiple times during a WEAKID treatment to examine its evolution during treatment (in mmHg).
Evolution of heart rate | This will be assessed during WEAKID treatment at t=0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Heart rate will be measured multiple times during a WEAKID treatment to examine its evolution during treatment (in beats per minute).
Evolution of body temperature | This will be assessed during WEAKID treatment at t=0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Body temperature will be measured multiple times during a WEAKID treatment to examine its evolution during treatment (in °C).
Evolution of oxygen saturation | This will be assessed during WEAKID treatment at t=0 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Oxygen saturation will be measured multiple times during a WEAKID treatment to examine its evolution during treatment (in %).
Ultrafiltration volume | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  For each WEAKID session, ultrafiltration volume will be determined (in mL).
Peak glucose concentration in the device effluent | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  For each WEAKID session, peak glucose concentration in the effluent of the device will be determined (in mmol/L).
Ultrafiltration efficiency | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  For each session, ultrafiltration efficiency (volume of osmotic water removal per gram absorbed glucose) will be determined (in mL/gram absorbed glucose).
Removal of urea by the WEAKID system | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The removal of urea (in mmol) by the WEAKID system will be determined for each WEAKID treatment
Removal of creatinine by the WEAKID system | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The removal of creatinine (in mmol) by the WEAKID system will be determined for each WEAKID treatment
Removal of phosphate by the WEAKID system | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The removal of phosphate (in mmol) by the WEAKID system will be determined for each WEAKID treatment
Removal of potassium by the WEAKID system | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The removal of potassium (in mmol) by the WEAKID system will be determined for each WEAKID treatment
Removal of beta-2 microglobulin by the WEAKID system | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The removal of beta-2 microglobulin (in mmol) by the WEAKID system will be determined for each WEAKID treatment
Mass transfer area coefficient of urea | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The mass transfer area coefficient (MTAC) for urea will be determined for each WEAKID treatment (in mL/min)
Mass transfer area coefficient of creatinine | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The mass transfer area coefficient (MTAC) for creatinine will be determined for each WEAKID treatment (in mL/min)
Mass transfer area coefficient of phosphate | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The mass transfer area coefficient (MTAC) for phosphate will be determined for each WEAKID treatment (in mL/min)
Mass transfer area coefficient of potassium | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The mass transfer area coefficient (MTAC) for potassium will be determined for each WEAKID treatment (in mL/min)
Mass transfer area coefficient of beta-2 microglobulin | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The mass transfer area coefficient (MTAC) for beta-2 microglobulin will be determined for each WEAKID treatment (in mL/min)
Plasma clearance of urea | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma clearance of urea will be determined for each WEAKID treatment (in mL/min)
Plasma clearance of creatinine | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma clearance of creatinine will be determined for each WEAKID treatment (in mL/min)
Plasma clearance of phosphate | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma clearance of phosphate will be determined for each WEAKID treatment (in mL/min)
Plasma clearance of potassium | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma clearance of potassium will be determined for each WEAKID treatment (in mL/min)
Plasma clearance of beta-2 microglobulin | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma clearance of beta-2 microglobulin will be determined for each WEAKID treatment (in mL/min)
The plasma reduction ratio of the protein-bound uremic toxin p-cresyl sulfate | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of p-cresyl sulfate will be calculated using the plasma concentrations before and after each WEAKID treatment.
The plasma reduction ratio of the protein-bound uremic toxin p-cresyl glucuronide | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of p-cresyl glucuronide will be calculated using the plasma concentrations before and after WEAKID treatment.
The plasma reduction ratio of the protein-bound uremic toxin indole acetic acid | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of indole acetic acid will be calculated using the plasma concentrations before and after WEAKID treatment.
The plasma reduction ratio of the protein-bound uremic toxin kynurenine | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of kynurenine will be calculated using the plasma concentrations before and after WEAKID treatment.
The plasma reduction ratio of the protein-bound uremic toxin kynurenic acid | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of kynurenic acid will be calculated using the plasma concentrations before and after WEAKID treatment.
The plasma reduction ratio of the protein-bound uremic toxin hippuric acid | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The plasma reduction ratio of hippuric acid will be calculated using the plasma concentrations before and after WEAKID treatment.
The release of base | This will be assessed for every WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  The release of base (in mmol) will be determined by calculating the sum of the release of bicarbonate (in mmol) and that of lactate (in mmol) for each WEAKID treatment
Evolution of plasma levels of urea | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Urea plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of creatinine | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Creatinine plasma levels (in micromol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of uric acid | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Uric acid plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of beta-2 microglobulin | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Beta-2 microglobulin plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of phosphate | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Phosphate plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of potassium | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Potassium plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of bicarbonate | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Bicarbonate plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of lactate | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Lactate plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of sodium | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Sodium plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of chloride | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Chloride plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of calcium | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Calcium plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of magnesium | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Magnesium plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of glucose | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Glucose plasma levels (in mmol/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of lactate dehydrogenase | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Lactate dehydrogenase plasma levels (in U/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of vitamin B12 | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Vitamin B12 plasma levels (in mg/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of albumin | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Albumin plasma levels (in g/L) will be determined before and after every WEAKID session.
Evolution of plasma leucocyte count | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Leucocyte count in plasma (in x10^9/L) will be determined before and after every WEAKID session.
Evolution of plasma thrombocyte count | These will be assessed before (at t=0 minutes) and after (at t=240 minutes or t=480 minutes for the 4-hour and 8-hour treatment, respectively) the WEAKID treatment throughout the study treatment period (2 weeks in total per participant)
  Thrombocyte count in plasma (in x10^9/L) will be determined before and after every WEAKID session.
Evolution of plasma levels of C-reactive protein (CRP) | This will be assessed before and after every series of three WEAKID treatment throughout the study treatment period (two times per week, two weeks in total per participant)
  CRP plasma levels (in mg/L) will be determined before and after every series of three WEAKID sessions.
Evolution of plasma levels of bilirubin | This will be assessed before and after every series of three WEAKID treatment throughout the study treatment period (two times per week, two weeks in total per participant)
  Bilirubin plasma levels (in umol/L) will be determined before and after every series of three WEAKID sessions.
Evolution of plasma levels of aspartate transaminase (ASAT) | This will be assessed before and after every series of three WEAKID treatment throughout the study treatment period (two times per week, two weeks in total per participant)
  ASAT plasma levels (in U/L) will be determined before and after every series of three WEAKID sessions.
Evolution of plasma levels of alanine aminotransferase (ALAT) | This will be assessed before and after every series of three WEAKID treatment throughout the study treatment period (two times per week, two weeks in total per participant)
  ALAT plasma levels (in U/L) will be determined before and after every series of three WEAKID sessions.
Evolution of sodium levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Sodium levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of chloride levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Chloride levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of calcium levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Calcium levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of magnesium levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Magnesium levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of bicarbonate levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Bicarbonate levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of lactate levels in dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Lactate levels (in mmol/L) will be determined in dialysate effluent at various timepoints during every WEAKID treatment.
Evolution of pH of dialysate effluent | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  pH of dialysate effluent will be determined at various timepoints during every WEAKID treatment.
Total number of device deficiencies and adverse device effects | This will be assessed through study completion (four weeks in total per participant)
  All device deficiencies (DDs) and adverse device effects (ADEs) will be reported and quantified.
Evolution of delta intraperitoneal pressure during WEAKID treatment | This will be assessed during WEAKID treatment at t=15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours (for 8-hour treatment), and 8 hours (for 8-hour treatment) throughout the study treatment period (2 weeks in total per participant)
  Delta intraperitoneal pressure will be calculated using the following formula:
  intraperitoneal pressure during WEAKID treatment (in mbar) - intraperitoneal pressure at t=0 (in mbar). Intraperitoneal pressure is determined using the pressure sensors of the WEAKID device.
Patient tolerance (abdominal discomfort) | This will be assessed at baseline, during every WEAKID treatment (at t = 0 minutes, 15 minutes, 1 hour, 2 hours, 4 hours, and 8 hours (for 8-hour treatment), and at the end of the study period (4 weeks in total per participant).
  Abdominal discomfort (scored using a numeric rating scale between 0-10) will be determined multiple times throughout the study period.
Evolution of uremic symptoms | This will be assessed at baseline and on the day of the last WEAKID treatment of each treatment week (three times during three weeks in total per participant).
  Uremic symptoms will be scored using the Dialysis Symptom Index questionnaire; this is a questionnaire consisting of thirty yes/no questions regarding whether participants have experienced a certain symptom during the last week. If the answer is yes, the participant will score how much they have felt burdened by this specific symptom during the last week on a Likert scale from 0-4; the higher the score, the more burdened the participant felt.

OTHER OUTCOMES:
Baseline characteristics | These will be assessed at baseline
  At baseline, demographical, clinical, and laboratory data will be collected. These include age, gender, body mass index, blood pressure, heart rate, oxygen saturation, body temperature, medication usage, medical history (including cause of kidney failure and comorbidity scored using the Charlsons' and Davies' indices, residual kidney function, renal clearance, renal weekly Kt/V, estimated glomerular filtration rate, and dialysis-related data (duration of dialysis, PD treatment modality and scheme, peritoneal catheter type, history of peritoneal catheter dysfunction or infection, dialysis adequacy, and peritoneal weekly Kt/V.
Peritoneal equilibrium tests | This will be assessed once at baseline and once the week after the last WEAKID treatment week (four weeks in total per participant).
  The standard peritoneal membrane analysis will be performed to determine the function of the peritoneal membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Karin GF Gerritsen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Università degli studi di Modena e Reggio Emilia (UNIMORE), Modena, Modena, Italy
- University Medical Center Utrecht (UMCU), Utrecht, Utrecht, Netherlands
- Hospital Universario La Paz (SERMAS), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will only be available to other researchers upon request and after approval of the Principal Investigator since the data is privacy-sensitive (pseudonymized) and commercially sensitive.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The following data will be shared (under restrictions if seen fit by the Principal Investigator) upon request:
  * The raw data
  * The study protocol describing the methods and materials
  * The script to process the data
  * The scripts leading to tables and figures in the publication
  * A codebook with explanations on the variable names
  * A 'read_me.txt' file with an overview of files included and their content and use.
  The time period will be determined on a case-by-case basis. A data sharing agreement outlining the terms of use for the receiving party will be drawn up before data is transferred.
Access Criteria: Data will be shared upon request after approval from the PI. The access criteria will be determined on a case-by-case basis.

REFERENCES:
- [Background] van Gelder MK, Ligabue G, Giovanella S, Bianchini E, Simonis F, Hazenbrink DHM, Joles JA, Bajo Rubio MA, Selgas R, Cappelli G, Gerritsen KGF. In vitro efficacy and safety of a system for sorbent-assisted peritoneal dialysis. Am J Physiol Renal Physiol. 2020 Aug 1;319(2):F162-F170. doi: 10.1152/ajprenal.00079.2020. Epub 2020 Jun 1. PMID 32475132
- [Background] van Gelder MK, de Vries JC, Simonis F, Monninkhof AS, Hazenbrink DHM, Ligabue G, Giovanella S, Joles JA, Verhaar MC, Bajo Rubio MA, Selgas R, Cappelli G, Gerritsen KGF. Evaluation of a system for sorbent-assisted peritoneal dialysis in a uremic pig model. Physiol Rep. 2020 Dec;8(23):e14593. doi: 10.14814/phy2.14593. PMID 33278069
- See also: Website regarding project CORDIAL — https://projectcordial.eu/en